CLINICAL TRIAL: NCT05071391
Title: Role of Autophagy and Inflammasome in the Pathophysiology of Obesity: Effect of Weight Loss and Potential Therapeutic Implications
Brief Title: Autophagy and Inflammasome in Obesity: Effect of Weight Loss and Potential Therapeutic Implications
Status: Completed | Type: Observational
Sponsor: Milagros Rocha Barajas (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Hospital Universitario Doctor Peset (Other)
Responsible Party: Sponsor-Investigator, Milagros Rocha Barajas, Senior Researcher, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Other Study IDs: PI16/00301
Record Dates: First submitted 2021-09-16; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Obesity
Keywords: bariatric surgery; autophagy; inflammasome; atherosclerosis; cardiovascular disease
MeSH Terms: conditions — Obesity; Atherosclerosis; Cardiovascular Diseases | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese: Obese patients undergoing Roux-en-Y gastric bypass
  Interventions: Procedure: Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass — Gastric bypass, also called Roux-en-Y gastric bypass, is a type of weight-loss surgery that involves creating a small pouch from the stomach and connecting the newly created pouch directly to the small intestine. After gastric bypass, swallowed food will go into this small pouch of stomach and then directly into the small intestine, thereby bypassing most of your stomach and the first section of your small intestine.
  Gastric bypass is one of the most commonly performed types of bariatric surgery. Gastric bypass is done when diet and exercise haven't worked or when you have serious health problems because of your weight.
  Other Names: RYGB

SUMMARY:
The main aim of this project is to determine the implication of autophagy and inflammasome in the pathogenesis of obesity and related comorbidities, and to explore in depth the mechanisms associated with the activation of immune cells leading early stages of the atherosclerotic process and metabolic disease. The hypothesis of the present study is that weight loss mediated by Roux-en-Y gastric bypass (RYGB) improves the protein expression of markers of autophagy and inflammation within immune cells. Moreover, the investigators will explore the association of these mechanisms with the mitochondrial function and dynamics, Endoplasmic Reticulum (ER) stress an intracellular nutritional status of leukocytes (measured by fluorescence microscopy and western blot). Further, the potential relationship between changes in the mentioned intracellular pathways and systemic pathological mechanisms including oxidative stress, inflammation and glucose and lipid metabolism will be explored. Hence, serum carbonylated proteins, myeloperoxidase (MPO) levels, antioxidant enzymatic activities including SOD (Superoxide dismutase) and catalase, circulating cytokines, and glucose and lipid metabolism parameters will be evaluated in a cohort of obese subjects before and 12 months after RYGB intervention.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 30 kg/m^2
* duration of obesity over 5 years

Exclusion Criteria:

* history of drug abuse
* pregnancy or lactation
* neoplastic disease
* severe renal/hepatic disease
* history of cardiovascular disease
* chronic inflammatory disease
* secondary cause for obesity (hypothyroidism, Cushing's syndrome)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with obesity prescribed bariatric surgery to treat their obesity and related comorbidities
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in the protein expression of autophagy markers in leukocytes 12 months after the RYGB intervention | 12 months
  Relative expression of intracellular proteins related autophagy/mitophagy mechanisms (Beclin 1, ATG5, LC3II/I, NRB1, PINK1, MIEAP) assessed by western blot and normalized to the loading control protein.
Changes in the relative protein expression of inflammatory mediators in leukocytes 12 months after the RYGB intervention | 12 months
  Relative expression of intracellular proteins related to inflammatory pathways (MCP1, NF-kB) assessed by western blot and normalized to the loading control protein.

SECONDARY OUTCOMES:
Changes in the protein expression of markers of mitochondrial dynamics and function in leukocytes 12 months after the RYGB intervention. | 12 months
  Relative expression of proteins related to mitochondrial dynamics and function (OPA1, FIS1, MFN1, DRP1, MFN2, OXPHOS Complex, MTTFA, PGC1α, NRF1, BNIP3) assessed by western blot and normalized to the loading control protein. Changes in mitochondrial membrane potential of leukocytes after the intervention assessed by fluorescence dye TMRM.
Changes in the protein expression of markers of nutrient sensing and ER stress in leukocytes 12 months after the RYGB intervention. | 12 months
  Relative expression of proteins related to nutritional status, metabolism and Endoplasmic Reticulum (ER) stress (AMPK, SIRT1, ATF6, CHOP) assessed by western blot and normalized to the loading control protein.
Changes in superoxide production 12 months after the RYGB intervention. | 12 months
  Evaluation of superoxide production in leukocytes by means of fluorescence dye (Relative Fluorescence Units) as contributor to pro-oxidant processes.
Changes in serum MPO levels 12 months after the RYGB intervention. | 12 months
  Evaluation of serum levels of the prooxidant MPO by immunoassay ELISA (ng/mL) as contributor to pro-oxidant and pro-inflammatory processes.
Changes in protein carbonylation in serum 12 months after the RYGB intervention. | 12 months
  Evaluation of carbonyl groups in serum proteins by means of immunoassay ELISA (nmol/mg protein) as a marker of systemic oxidative damage.
Changes in serum SOD enzymatic activity 12 months after the RYGB intervention. | 12 months
  Evaluation of SOD enzymatic activity in serum (nmol/min/mL) as part of the systemic antioxidant defense system.
Changes in serum catalase enzymatic activity 12 months after the RYGB intervention. | 12 months
  Evaluation of catalase enzymatic activity in serum (nmol/min/mL) as part of the systemic antioxidant defense system.
Effect of the RYGB on body weight | 12 months
  Changes in the body weight (kg) of patients 12 months after the RYGB intervention determined with an electronic scale
Effect of the RYGB on Body Mass Index (BMI) | 12 months
  Changes in the BMI (kg/m^2) of patients 12 months after the RYGB intervention, measure by the formula: weight (kg) / [height (m)]^2
Effect of the RYGB on blood pressure | 12 months
  Changes in Systolic/Diastolic Blood Pressure levels (SBP/DBP) (mmHg) measured with a sphygmomanometer
Effect of the RYGB on fasting Glucose levels | 12 months
  Changes in fasting Glucose (mg/dL) of patients 12 months after the RYGB intervention, as a marker of glucose metabolism
Effect of the RYGB on fasting Insulin levels | 12 months
  Changes in fasting Insulin (μU/mL) of patients 12 months after the RYGB intervention, as a marker of glucose metabolism
Effect of the RYGB on Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) Index | 12 months
  Changes in HOMA-IR Index of patients 12 months after the RYGB intervention, measured with the formula: [Fasting Glucose (mg/dL) x Fasting Insulin (μU/mL)]/405, as a marker of glucose metabolism
Effect of the RYGB on glycated hemoglobin (HbA1c) | 12 months
  Changes in HbA1c (%) of patients 12 months after the RYGB intervention, as a marker of glucose metabolism
Effect of the RYGB on Total Cholesterol (TC) | 12 months
  Changes in TC (mg/dL) of patients 12 months after the RYGB intervention, as a marker of the lipid profile
Effect of the RYGB on High Density Lipoprotein Cholesterol (HDLc) levels | 12 months
  Changes in HDLc (mg/dL) of patients 12 months after the RYGB intervention, as a marker of the lipid profile
Effect of the RYGB on Low Density Lipoprotein Cholesterol (LDLc) levels | 12 months
  Changes in LDLc (mg/dL) of patients 12 months after the RYGB intervention, as a marker of the lipid profile
Effect of the RYGB on Triglyceride (TG) levels | 12 months
  Changes in TG (mg/dL) of patients 12 months after the RYGB intervention, as a marker of the lipid profile
Effect of the RYGB on high sensitivity C-Reactive Protein (hsCRP) levels | 12 months
  Changes in hsCRP (mg/L) of patients 12 months after the RYGB intervention, as a marker of systemic inflammation
Effect of the RYGB on Interleukin-6 (IL6) levels | 12 months
  Changes in IL6 (pg/mL) of patients 12 months after the RYGB intervention, as a marker of systemic inflammation
Effect of the RYGB on Interleukin-1 β (IL1β) levels | 12 months
  Changes in IL1β (pg/mL) of patients 12 months after the RYGB intervention, as a marker of systemic inflammation
Remission rate for pathologies related to metabolic syndrome 12 months after RYGB intervention | 12 months
  Percentage of cases of remission for hypertension, hyperlipidemia and type 2 diabetes (T2D) after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Milagros Rocha Barajas, PhD, Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Locations (1):
- Hospital Universitario Doctor Peset, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No